CLINICAL TRIAL: NCT02278094
Title: A Randomized Controlled Study to Examine the Effect of Home-based Recovery Activity in Moderate to Severe Obstructive Sleep Apnea Syndrome Patients
Brief Title: The Influences of Intervention With Home-based Recovery Activity in Obstructive Sleep Apnea Syndrome
Acronym: OSAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: --/A-ER-103-168
Record Dates: First submitted 2014-09-28; First posted 2014-10-29 (Estimated); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Obstructive Sleep Apnea
Keywords: OSAS; Adult; Home-based; Genioglossus; Inspiratory muscle; Exercise
MeSH Terms: conditions — Sleep Apnea, Obstructive; Motor Activity | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental group (Experimental): Subjects will be in random cluster assign to walking exercise (WE), Threshold Inspiratory Muscle Trainer (TIMT) and Tongue Muscle Trainer (TMT) treatment groups.
  Interventions: Device: Tongue Muscle Trainer (TMT); Device: Threshold Inspiratory Muscle Trainer (TIMT); Procedure: Walking Exercise
- Control group (Active Comparator): Up to 95% of OSAS cases are treated with continuous positive airway pressure (CPAP), CPAP treatment group will be the control group.
  Interventions: Device: Continuous Positive Airway Pressure (CPAP)

INTERVENTIONS:
Device: Tongue Muscle Trainer (TMT) — Subject will be instructed to compress the Iowa Oral Performance Instrument (IOPI) IOPI's bulb using tongue in three directions (anterior and both lateral sides). Then, hold 30-35 seconds each time. Subjects will be encouraged to do 60 minutes of exercise daily then continue three to five times a week for a total of 3 months.
  Arms: Experimental group
Device: Threshold Inspiratory Muscle Trainer (TIMT) — Resistance of the TIMT devices will be set from 30% of the maximum inspiratory pressure. Nose clip follow by normal breathing. Seal the mouth to the device's mouth piece then inhale through the device. Subjects will be encouraged to do 60 minutes of exercise daily then continue three to five times a week for a total of 3 months.
  Arms: Experimental group
Procedure: Walking Exercise — Subjects will be encouraged to perform walking exercise in the field 10000 steps/ 60 minutes daily then continue three to five times a week during first months. Followed by 12500 steps and 15000steps per day during the second and third months.
  Arms: Experimental group
Device: Continuous Positive Airway Pressure (CPAP) — CPAP regular therapy per day (use ≥ 4 h/day) then continue three to five times a week for a total of 3 months.
  Arms: Control group

SUMMARY:
Background: OSAS is a type of sleep disorder characterized by intermittent, partial or complete upper airway (UA) collapse, seriously impacting sleep apnea and respiratory insufficiency. The major upper airway dilator muscle (genioglossus) is more active during periods of stable breathing compared with periods of cyclical breathing when obstructive apneas occurred. UA muscle strength is linearly related to the inspiratory pump muscle strength. The ratios of UA muscle strength (tongue protrusion, TP) and inspiratory pump muscle strength (PImax) were not different between individuals with and without OSAS. However, a highly wakeful ratio of TP force to PImax appears to be associated with a reduced propensity to moderate-to-severe OSAS. Up to 95% of OSAS cases are treated with continuous positive airway pressure (CPAP), which is the most effective, commonly used, and low-risk treatment method. However, patients using CPAP therapy could face ongoing difficulties. Aims: To evaluate the effects of home-based exercise for patients with moderate to severe OSAS. This study was a randomized clinical trial conducted at three different intervention protocols as experimental groups. We will use cluster random sampling assign to each group. CPAP treatment group will be the control group. Methods: Subject above 20 years old will be diagnosed to moderate and severe OSAS. Subjects will be assign to walking exercise (WE), Threshold Inspiratory Muscle Trainer (TIMT) and Tongue Muscle Trainer (TMT) treatment groups. We will compare the Polysomnography (PSG) data, Epworth Sleepiness scale (ESS), World Health Organization Quality of Life( WHOQOL) questionnaire is a shorter version of the original instrument (WHOQOL-BREF), 6-minute walking test (6MWD), rate of perceived exertion scale (RPE), flow-volume loop (FV-Loop), tongue and grasp muscle strength, anthropometric data and daily note at baseline, 3 months (end-of-intervention) and 6 months (post intervention follow-up) in patients with moderate to severe OSAS. They will undergo three months of the home-based exercises. Patients will be followed up with weekly telephone calls and be interviewed monthly. Expected results: By using the WE, TIMT and TMT therapies, the airway collapse during sleep will be prevented when the whole body muscle strength, inspiratory pump muscle strength and tongue muscle strength are enhanced.

DETAILED DESCRIPTION:
Obstructive sleep apnea syndrome (OSAS) is a common form of sleep-disordered breathing (SDB) characterized by repetitive episodes of cessation of breathing during sleep due to upper airway collapse. It causes sleep fragmentation, disabling daytime sleepiness, impaired cognitive function and poor quality of life. In addition, OSAS is associated with non-fatal and fatal cardiovascular consequences including sudden death as well as to an increased risk of road traffic accidents. OSAS is a common disease, affecting approximately 2% of women and 4% of men residing in Western communities.

Risk factors for OSAS include obesity, aging, particularly males, abnormal craniofacial morphology, nasal obstruction, and genetic factors. OSAS is associated with several cardiovascular consequences and social consequences such as motor vehicle accidents, impaired cognitive performance, and depression. Various epidemiologic studies have shown an association between OSAS and hypertension. In a cross-sectional study, OSAS was associated with increased prevalence of self-reported heart failures and strokes. OSAS has been shown to be independently associated with coronary artery disease after adjustment for traditionally considered risk factors.

According to the American Medical Association in 2013, obstructive sleep apnea syndrome (OSAS) is a common disorder that affects everyone in all ages, especially middle-aged and elderly people. In fact, evidence showed that OSAS rates had been increasing due to the escalation of obesity rates. Thus, the goal of the OSAS treatment is to alleviate the airway obstruction during sleep. The standard first-line OSAS treatment involves continuous positive airway pressure (CPAP) devices, which deliver compressed air into the airway in order to stay open. In most cases, many patients cannot tolerate CPAP and often are unable to adhere to the instructions for many reasons. Patients began to feel discomfort and claustrophobic as well as skin irritation and noise. Although small studies lack data of other OSAS treatments, this case resulted in insufficient evidence to determine the efficacy of these strategies. In regards to limited data, the evidence is not yet resolved on the effectiveness of the treatment. There is very limited evidence on the clinical outcomes of the OSAS intervention, and most of the data focus on immediate results that are exceedingly direct and provide no long-term benefits. Likewise, evidence in evaluating the relative efficacy of weight loss, oronasopharyngeal exercise and tongue retraining device interventions for OSAS treatment was insufficient. Low-quality evidence indicated that the above interventions improved sleep measures and should be recommended for patients with OSAS.

Purpose:

The aim of the study was to assess the effect of PSG data, Epworth Sleepiness scale (ESS), WHOQOL-BREF questionnaire (EQ-5D), 6-minute walking test (6MWD), rate of perceived exertion scale (RPE), flow-volume loop (FV-Loop), tongue and grasp muscle strengths, anthropometric data and daily note record between two groups (control group: CPAP therapy and experimental group: subgroup have WE, TIMT and TMT therapies) patients with moderate to severe obstructive sleep apnea syndrome (OSAS).

Hypothesis:

The investigators hypothesize that more moderate to severe obstructive sleep apnea syndrome patients in a home-based recovery activity intervention program will have improved PSG data, quality of life, exercise ability, pulmonary function, muscle strength, anthropometric data and daily note record than patients receiving CPAP alone.

ELIGIBILITY:
Inclusion Criteria:

* Mean aged ≥20 years old,
* Good general health (stability of clinic state)
* Epworth Sleepiness Scale ≥ 10
* PSG for discriminate moderate to severe subjects (AHI≧15 h-1)
* Presence of excessive daytime somnolence (EDS)
* From the community and hospital

Exclusion Criteria:

* Inability to exercise
* Exercise-induced myocardial ischemia
* Chronic pulmonary disease
* Stroke
* Peripheral arterial disease
* Severe psychiatric disorder (e.g. bipolar disorder, schizophrenia)
* Tensile hypertrophy
* Pregnancy
* Alcoholism (≥ 50 gm per day)
* Active or uncontrolled chronic medical condition (e.g., cardio-respiratory disease, diabetes mellitus, endocrine disorders, stroke, abnormal pulmonary function, morbid obesity, renal disease, hypertension (i.e., >159/99 mm Hg), myopathy, neurologic illness, recent infection , and recent (< 3 months) myocardial infarction, or angina).

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2014-09; Primary Completion 2020-05 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Polysomnography(PSG) data in the scoring of apnea-hypopnea index (AHI), sleep stages and respiratory events. | Baseline, post-intervention (3 months) and post-intervention follow (6 months after ceasation of intervention)
  The sleep efficacy will be calculated by the parameters of PSG.

SECONDARY OUTCOMES:
Epworth Sleepiness Score (ESS) | Baseline, post-intervention (3 months) and post-intervention follow (6 months after ceasation of intervention)
  The Epworth Sleepiness Scale (ESS) is a questionnaire for assessing daytime sleepiness.
WHOQOL-BREF(EQ-5D) questionnaire | Baseline , post-intervention (3 months) and post-intervention follow (6 months after ceasation of intervention)
  The utility value of the QOL for patients on Prolonged Mechanical Ventilation (PMV) was estimated using the EuroQol five-dimensional (EQ-5D) questionnaire, which is a generic preference-based instrument.
6MWD( = 6MWT) | Baseline, post-intervention (3 months) and post-intervention follow (6 months after ceasation of intervention)
  The 6-min walk test (6MWT), which is a cheap and simple examination to perform, is now regarded as a standard tool to measure submaximal exercise capacity in patients with cardiopulmonary disease.
RPE | Baseline, post-intervention (3 months) and post-intervention follow (6 months after ceasation of intervention)
  Ratings of perceived exertion (or "effort and exertion") are important complements toward physiological measurements. Of all the single indicators of the degree of physical strain, perceived exertion is one of the most directive measures.
Flow-volume loop (FV-Loop) | Baseline, post-intervention (3 months) and post-intervention follow (6 months after ceasation of intervention)
  The flow-volume curve is important and may help interpret pulmonary symptoms or upper airway diseases.
Tongue Muscle Strength | Baseline, post-intervention (3 months) and post-intervention follow (6 months after ceasation of intervention)
  The measurement of tongue strength contributes to the study of oro-facial physiology.
Anthropometric data | Baseline, post-intervention (3 months) and post-intervention follow (6 months after ceasation of intervention)
  Anthropometric measurements including height, weight, and circumference measurements were obtained before and after the study.

CONTACTS AND LOCATIONS:
Overall Officials: Hung Ching-Hsia, PT, Principal Investigator — National Cheng Kung University
Locations (1):
- Tainan Hospital (Ministry of Health and Welfare), Tainan, Taiwan